CLINICAL TRIAL: NCT03310411
Title: A Randomized, Double-Blind, Four-Period, Crossover Study to Evaluate the Cardiovascular Effect of Single Oral Doses of Lasmiditan When Coadministered With Single Oral Doses of Sumatriptan in Healthy Subjects
Brief Title: A Study of Lasmiditan When Given With Sumatriptan in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16926; H8H-MC-LAHU (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2018-01

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lasmiditan + Sumatriptan (A) (Experimental): Single oral dose of 200 milligram (mg) lasmiditan tablet and single oral dose of 100 mg sumatriptan tablet in one of four treatment periods.
  Interventions: Drug: Lasmiditan; Drug: Sumatriptan
- Lasmiditan + Placebo (B) (Experimental): Single oral dose of 200 mg lasmiditan tablet and single oral dose of placebo tablet in one of four treatment periods.
  Interventions: Drug: Lasmiditan; Drug: Placebo for Sumatriptan
- Sumatriptan + Placebo (C) (Active Comparator): Single oral dose of 100 mg sumatriptan tablet and single oral dose of placebo tablet in one of four treatment periods.
  Interventions: Drug: Sumatriptan; Drug: Placebo for Lasmiditan
- Placebo + Placebo (D) (Placebo Comparator): Oral doses of placebo tablets in one of four treatment periods.
  Interventions: Drug: Placebo for Lasmiditan; Drug: Placebo for Sumatriptan

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144
  Arms: Lasmiditan + Placebo (B); Lasmiditan + Sumatriptan (A)
Drug: Sumatriptan — Administered orally
  Arms: Lasmiditan + Sumatriptan (A); Sumatriptan + Placebo (C)
Drug: Placebo for Lasmiditan — Administered orally
  Arms: Placebo + Placebo (D); Sumatriptan + Placebo (C)
Drug: Placebo for Sumatriptan — Administered orally
  Arms: Lasmiditan + Placebo (B); Placebo + Placebo (D)

SUMMARY:
The purpose of this study is to assess whether taking lasmiditan and sumatriptan together will have any additional effects on heart rate and blood pressure compared to taking lasmiditan and sumatriptan individually. This study will also look at the amount of study drug that gets into the blood stream and how long it takes the body to get rid of it when these two drugs are taken together.

This study will last about 21 days, not including the screening. Participants will spend 16 days/15 nights in the clinical research unit (CRU) followed by follow-up. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Have a body mass index of 19.0 to 35.0 kilograms per meter squared (kg/m²) inclusive

Exclusion Criteria:

* Have known allergies to Lasmiditan, Sumatriptan, related compounds, or any components of the formulations of Lasmiditan and Sumatriptan
* Have a history of, or electrocardiogram (ECG) findings of, clinically significant bradycardia, heart block, tachy or brady arrhythmias
* Have a history, signs, or symptoms of arrhythmia or Wolff Parkinson White syndrome that could affect the participant's safety
* Have an estimated glomerular filtration rate (eGFR) of less than (<) 60 milliliter per minute (mL/min) per 1.73 m²
* Have a resting systolic blood pressure (SBP) greater than (>) 135 millimeters of mercury (mmHg) and diastolic blood pressure (DBP) >85 mmHg at screening
* Have a supine pulse rate (PR) of <50 or >90 beats per minute (bpm) at screening
* Have a history, signs, or symptoms of vasospastic coronary artery disease
* Have known or ongoing neuropsychiatric disorders (for example, manic depressive illness, schizophrenia, depression) considered as clinically significant by the investigator
* Use of monoamine oxidase-A inhibitors and other drugs associated with serotonin within the 3 months prior to the first dosing occasion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Daytona Beach, Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover study with four periods. Participants were randomized to one of four treatment (Treatment A: 200 milligram (mg) lasmiditan + 100mg sumatriptan, Treatment B: 200mg lasmiditan + placebo, Treatment C: 100mg sumatriptan + placebo, Treatment D: placebo + placebo) period sequences. There was a washout of at least 4 days between each dosing day.
Groups:
- Sequence 1: Participants received single oral dose of Lasmiditan, sumatriptan and placebo tablets on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 200 mg Lasmiditan + 100 mg sumatriptan, Period 2: 200 mg Lasmiditan + placebo Period 3: 100 mg Sumatriptan + placebo Period 4: Placebo + placebo
- Sequence 2: Participants received single oral dose of Lasmiditan, sumatriptan and placebo tablets on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 200 mg Lasmiditan + placebo Period 2: 100 mg Sumatriptan + placebo Period 3: Placebo + placebo Period 4: 200 mg Lasmiditan + 100 mg sumatriptan
- Sequence 3: Participants received single oral dose of Lasmiditan, sumatriptan and placebo tablets on day 1 of each treatment period as per the below dosing sequence.
  Period 1: 100 mg Sumatriptan + placebo Period 2: Placebo + placebo Period 3: 200 mg Lasmiditan + 100 mg sumatriptan Period 4: 200 mg Lasmiditan + placebo
- Sequence 4: Participants received single oral dose of Lasmiditan, sumatriptan and placebo tablets on day 1 of each treatment period as per the below dosing sequence.
  Period 1: Placebo + placebo Period 2: 200 mg Lasmiditan + 100 mg sumatriptan Period 3: 200 mg Lasmiditan + placebo Period 4: 100 mg Sumatriptan + placebo
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 10 | 10 | 10 | 10
Received at Least 1 Dose of Study Drug | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 10 | 10 | 10 | 9
Completed | 10 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 10 | 10 | 10 | 9
Completed | 10 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Period Title: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 10 | 10 | 10 | 9
Completed | 10 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Overall: Participants received single oral dose of 200 mg lasmiditan, 100 mg sumatriptan, 200 mg lasmiditan + 100 mg sumatriptan or placebo tablets on Day 1 of each treatment period according to their assigned treatment sequence.
Arm/Group | Overall
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics (PD): Change From Baseline in Mean 24-hour Systolic Blood Pressure (SBP)
Description: Systolic Blood Pressure (SBP) was measured by using a 24-hour Ambulatory Blood Pressure Monitoring (ABPM) device attached to the participant's nondominant arm. Ambulatory blood pressure measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least squares (LS) mean peak changes from baseline were calculated using a linear mixed-effects model with baseline, treatment, period, and sequence as fixed effects and participant as a random effect.
Time Frame: Baseline (Day 1), Day 2
Population: All enrolled participants who received at least one dose of study drug with evaluable blood pressure data.
Measure: Least Squares Mean (90% Confidence Interval); unit: Millimeters of mercury (mmHg)
Groups:
- 200 mg Lasmiditan + 100 mg Sumatriptan (A):: Participants received single oral dose of 200 mg lasmiditan tablet and single oral dose of 100 mg Sumatriptan tablet on day1.
- 200 mg Lasmiditan + Placebo (B): Participants received single oral dose of 200 mg lasmiditan tablet and single oral dose of placebo tablet on day 1.
- 100 mg Sumatriptan + Placebo (C): Participants received single oral dose of 100mg sumatriptan tablet and single oral dose of placebo tablet on day 1.
- Placebo + Placebo (D): Participants received single oral dose of placebo for lasmiditan tablet and single oral dose of placebo for sumatriptan tablet on day 1.
Arm/Group | 200 mg Lasmiditan + 100 mg Sumatriptan (A): | 200 mg Lasmiditan + Placebo (B) | 100 mg Sumatriptan + Placebo (C) | Placebo + Placebo (D)
Number analyzed (Participants) | 39 | 38 | 39 | 39
Millimeters of mercury (mmHg) | 13.81 [11.83 to 15.79] | 12.17 [10.47 to 13.87] | 13.63 [11.65 to 15.61] | 11.42 [9.74 to 13.09]

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Lasmiditan and Sumatriptan
Description: PK: Cmax of Lasmiditan and Sumatriptan was evaluated.
Time Frame: Lasmiditan: Predose, 0.5, 1, 1.5,2, 2.5, 3, 4, 6, 8, 12 , 24 ,36 and 48 hours(h) postdose; Sumatriptan: Predose, 0.5, 1, 1.5,2, 2.5, 3, 4, 6, 8, 12 and 24 h postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 200 mg Lasmiditan + 100 mg Sumatriptan (A):Analyte: Lasmiditan; 200 mg Lasmiditan +100 mg Sumatriptan (A):Analyte: Sumatriptan: Participants received single oral dose of 200 mg lasmiditan tablet and single oral dose of 100 mg sumatriptan tablet on day 1.
- 200 mg Lasmiditan + Placebo (B): Analyte: Lasmiditan: Participants received single oral dose of 200 mg lasmiditan tablet and single oral dose of placebo tablet on day 1.
- 100 mg Sumatriptan + Placebo (C): Analyte: Sumatriptan: Participants received single oral dose of 100mg sumatriptan tablet and single oral dose of placebo tablet on day 1.
Arm/Group | 200 mg Lasmiditan + 100 mg Sumatriptan (A):Analyte: Lasmiditan | 200 mg Lasmiditan + Placebo (B): Analyte: Lasmiditan | 200 mg Lasmiditan +100 mg Sumatriptan (A):Analyte: Sumatriptan | 100 mg Sumatriptan + Placebo (C): Analyte: Sumatriptan
Number analyzed (Participants) | 39 | 39 | 39 | 38
nanogram per milliliter (ng/mL) | 304 (39) | 328 (32) | 56.8 (36) | 50.7 (42)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0 ∞]) of Lasmiditan and Sumatriptan
Description: PK: AUC(0 ∞) of Lasmiditan and Sumatriptan was evaluated.
Time Frame: Lasmiditan: Predose, 0.5, 1, 1.5,2, 2.5, 3, 4, 6, 8, 12, 24 ,36 and 48 h postdose; Sumatriptan: Predose, 0.5, 1, 1.5,2, 2.5, 3, 4, 6, 8, 12 and 24 h postdose
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- 200mg Lasmiditan + 100mg Sumatriptan (A): Analyte: Lasmiditan; 200 mg Lasmiditan +100 mg Sumatriptan (A):Analyte: Sumatriptan: Participants received single oral dose of 200 mg lasmiditan tablet and single oral dose of 100 mg sumatriptan tablet on day 1.
- 100 mg Sumatriptan + Placebo (C): Analyte: Sumatriptan: Participants received single oral dose of 100 mg sumatriptan tablet and single oral dose of placebo tablet on day 1.
Arm/Group | 200mg Lasmiditan + 100mg Sumatriptan (A): Analyte: Lasmiditan | 200 mg Lasmiditan + Placebo (B): Analyte: Lasmiditan | 200 mg Lasmiditan +100 mg Sumatriptan (A):Analyte: Sumatriptan | 100 mg Sumatriptan + Placebo (C): Analyte: Sumatriptan
Number analyzed (Participants) | 39 | 39 | 39 | 38
nanogram*hour per milliliter (ng*hr/mL) | 2110 (37) | 2170 (33) | 253 (28) | 240 (29)

ADVERSE EVENTS:
Time Frame: Up To 36 Days
Description: All enrolled participants who received at least one dose of study drug and had at least one post-dose safety assessment.
Groups:
- 200 mg Lasmiditan + 100 mg Sumatriptan (A): Participants received single oral dose of 200 mg lasmiditan tablet and single oral dose of 100 mg sumatriptan tablet on day 1.
- 200 mg Lasmiditan + Placebo (B): Participants received single oral dose of 200mg lasmiditan tablet and single oral dose of placebo tablet on day 1.
Arm/Group | 200 mg Lasmiditan + 100 mg Sumatriptan (A) | 200 mg Lasmiditan + Placebo (B) | 100 mg Sumatriptan + Placebo (C) | Placebo + Placebo (D)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 4/39 | 7/39 | 3/39 | 1/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Lasmiditan + 100 mg Sumatriptan (A) (N=39) | 200 mg Lasmiditan + Placebo (B) (N=39) | 100 mg Sumatriptan + Placebo (C) (N=39) | Placebo + Placebo (D) (N=40)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 5 (5) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.

DOCUMENTS (2):
  • Study Protocol (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT03310411/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03310411/SAP_001.pdf